CLINICAL TRIAL: NCT00832156
Title: Application of Cultured Autologous Keratinocytes in Combination With a Meshed Split Skin Autograft for Burn Wound Healing
Brief Title: Application of Cultured Autologous Keratinocytes for Burn Wound Healing
Acronym: KC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBS 07.116 KC; NL19048.000.07
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2014-06

CONDITIONS: Burns
Keywords: Burns; Cultured autologous keratinocytes; Wound healing; Wound closure; Scar quality
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): wound 1: the placement of keratinocytes onto a collagen/elastin support after the application of the meshed split skin autograft.
  Interventions: Biological: Cultured autologous keratinocytes
- 2 (Other): control wound site; application of mesh graft alone
  Interventions: Biological: Cultured autologous keratinocytes

INTERVENTIONS:
Biological: Cultured autologous keratinocytes — The experimental wound site will be covered with cultured keratinocytes on a collagen/elastin carrier after the application of a meshed split skin autograft. The control wound site will be covered with a meshed split skin autograft alone.
  Other Names: Cultured keratinocytes

SUMMARY:
In this study the treatment of full thickness burn wounds with cultured autologous keratinocytes in combination with meshed split skin autograft versus meshed split skin graft alone will be compared. It is expected that the application of cultured autologous keratinocytes in combination with a meshed split skin autograft will improve wound healing and scar formation.

DETAILED DESCRIPTION:
The standard treatment for extensive burn wounds is transplantation with meshed split skin graft. Disadvantages of this treatment are that healing of large full thickness burn wounds is still accompanied by scar formation. Even standard treatment, transplantation with a (meshed) split skin autograft, does not result in satisfactory functional and cosmetic appearance of the healed wound. Due to limited available donor sites meshes needs to be enlarged. Bigger enlargements of meshes give more scarring and mesh pattern are still visible in scars, probably because wound closure still needs several weeks. Application of cultured autologous keratinocytes may enhance wound closure and improve outcome of healing.

Primary objective: Does the application of cultured autologous keratinocytes on deep burn wounds accelerate wound closure Secondary objectives: Does the application of cultured autologous keratinocytes on deep burn wounds improve scar quality with respect to scar elasticity, colour/pigmentation and/or smoothness after 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Competent and temporarily incompetent patients 18 years of age or older with acute burn wounds that require widely meshed skin grafting, which do not need immediate excision
* Minimal study wound area 100 cm2
* Maximal study wound area 300 cm2
* Maximal TBSA 30% full thickness wounds
* Informed consent

Exclusion Criteria:

* Immunocompromised patients
* Infected wounds
* Use of high doses of (.20mg/pd) corticosteroids and/or cytostatica
* Known penicillin allergy
* Conditions where the patient is non compliant as judged by a medical specialist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Primary end point is the percentage of wound closure. | 7 days

SECONDARY OUTCOMES:
Secondary objective is scar quality (i.e. subjective scar assessment, scar elasticity, colour and pigmentation of the scar and smoothness of the scar surface). | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: E Middelkoop, Prof, Study Director — Association of Dutch Burn Centers
Locations (1):
- Red Cross Hospital, Beverwijk, North Holland, Netherlands